CLINICAL TRIAL: NCT00861874
Title: A Phase I Study of Decitabine in Combination With Escalating Doses of Rapamycin in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: A Study of Decitabine in Combination With Escalating Doses of Rapamycin in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jane Liesveld, Professor of Medicine, Hematology and Bone Marrow Transplant, University of Rochester
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26037
Record Dates: First submitted 2009-03-12; First posted 2009-03-16 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Decitabine; Drug: Rapamycin

INTERVENTIONS:
Drug: Decitabine — 20 mg/m2 IV, Days 1-5
Drug: Rapamycin — Dose level 1 = 2mg/daily, Dose level 2 = 4mg/daily, Dose level 3 = 6mg/daily. Oral, Days 6-26

SUMMARY:
The purpose of this study is to determine the safety and feasibility of the combination of decitabine given at a fixed dose with escalating doses of rapamycin in patients with relapsed or refractory acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Diagnosis of AML according to WHO criteria except acute promyelocytic leukemia AND
* Refractory AML defined as a failure to achieve CR after 2 cycles of induction chemotherapy or persistence of > 40% bone marrow blasts after one cycle of chemotherapy induction OR
* Relapsed AML defined as any evidence of disease recurrence within 12 months of achieving first CR OR
* Relapsed AML after stem cell transplantation 100 days must have elapsed between transplant and emergence of recurrent AML
* ECOG performance status <3 (Appendix 1)

Exclusion Criteria:

* Abnormal renal function as evidenced by a calculated creatinine clearance ≤ 30ml/min (Cockcroft-Gault formula (Appendix 2)
* Abnormal liver function: Bilirubin >2.0 mg/dl, transaminase more than 2.5x the upper limits of normal
* Active systemic infection
* Known chronic liver disease
* Known diagnosis of human immunodeficiency virus infection (HIV)
* Patients who are post-allogeneic transplantation should not have active GVHD greater than grade 1 of skin
* Pregnant or breast feeding female subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of chemotherapy with the drug decitabine combined with rapamycin to determine the highest dose of rapamycin that can be given in combination with decitabine. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jane Liesveld, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Liesveld JL, O'Dwyer K, Walker A, Becker MW, Ifthikharuddin JJ, Mulford D, Chen R, Bechelli J, Rosell K, Minhajuddin M, Jordan CT, Phillips GL 2nd. A phase I study of decitabine and rapamycin in relapsed/refractory AML. Leuk Res. 2013 Dec;37(12):1622-7. doi: 10.1016/j.leukres.2013.09.002. Epub 2013 Sep 8. PMID 24138944